CLINICAL TRIAL: NCT01159392
Title: Effects of Recruitment Maneuvers in Patients With Acute Brain Injury and Acute Lung Injury
Brief Title: Alveolar Recruitment in Brain Injury
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Elizabeth Zavala, Hospital Clinic
Other Study IDs: RM-0152; FIS-0152 (Other Grant/Funding Number: Fondo de Investigaciones Sanitarias)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2001-02

CONDITIONS: Brain Injury; Acute Lung Injury
Keywords: brain injury; mechanical ventilation; acute lung injury; lung recruitment
MeSH Terms: conditions — Brain Injuries; Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain injury plus acute lung injury: Patients with severe brain injury (Glasgow coma score<13) with acute lung injury (PaO2/FiO2 <300 mmHg)

SUMMARY:
Development of acute lung injury (ALI) and acute respiratory distress syndrome (ARDS) in patients with severe brain injury has been associated with poor outcome. The application of lung recruitment maneuvers (RM) for a short period of time to open collapsed alveoli and reverse hypoxemia in early ARDS has been recommended. However, little is known about the cerebral and vascular effects of RM in brain injury patients with ALI/ARDS. The aim of this study is to assess the effects of a single standardized RM on oxygenation and on systemic and cerebral hemodynamics in severe brain injury patients with ALI/ARDS.

DETAILED DESCRIPTION:
Patients with severe brain injury comprise a significant portion of admissions to critical care units. These patients are unable to adequately protect their airways and are usually intubated and mechanically ventilated. The goal of mechanical ventilation in patients with brain injury is to optimize blood gas exchange while minimizing intrathoracic pressure to avoid interference with cerebral venous drainage.Over the last 20 years, a plethora of experimental and clinical data have shown that mechanical ventilation can cause or aggravate lung damage in patients with acute lung injury (ALI) and the acute respiratory distress syndrome (ARDS). The aim of this pilot study was to assess the effects of a single standardized recruitment maneuver (RM) on oxygenation and on systemic and cerebral hemodynamics in severe brain injury patients with ALI/ARDS.

Only patients with brain injury, as defined by a Glasgow Coma Score <13, admitted into the Trauma and Surgical intensive care unit (ICU) will be studied.

After obtaining informed consent, a RM will be performed by switching the ventilator from assist/control ventilation to continuous positive airway pressure (CPAP) and applying a pressure of 40 cmH2O for 40 sec (11). After the RM, patients have been ventilated in pressure control ventilation and PEEP will be gradually reduced in decremental steps every 3 respiratory cycles starting with PEEP at 30 cm H2O, maintaining a maximum peak pressure of 40 cmH2O during this procedure until pre-RM PEEP levels are achieved. The RM will be discontinued if any of the following changes developed during the procedure: (i) ≥20% changes in baseline systemic blood pressure, (ii) ICP ≥20 mmHg, or (iii) SaO2 ≤90%. After the RM is performed, respiratory mechanics, arterial and SjO2 blood samples and systemic and cerebral hemodynamics will be obtained at 30 min and 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain injury who met the ALI/ARDS criteria within 72 hours after ICU admission

Exclusion Criteria:

* <18 years of age
* Cardiogenic edema
* Hemodynamic instability
* Intracranial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain injury (Glasgow Coma Score<13) admitted into the Trauma and Surgical Intensive care unit (ICU) at the Hospital Clinic, Barcelona.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2001-02; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
arterial oxygenation | 8 hours
  Arterial oxygenation was expressed as PaO2/FiO2 ratio

SECONDARY OUTCOMES:
cerebral hemodynamics | 8 hours
  Cerebral hemodynamics will be assessed by cerebral perfusion pressure and intracranial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Zavala, MD, PhD, Principal Investigator — Hospital Clinic, Barcelona, Spain
Locations (1):
- Trauma and Surgical ICU, Hospital Clinic, Barcelona, Spain